CLINICAL TRIAL: NCT01969201
Title: Randomised Clinical Trial Comparing Highly Purified FSH Formulation (Fostimon®) and Recombinant FSH (Gonal-F®) in GnRH-antagonist Controlled Ovarian Hyperstimulation Cycles.
Brief Title: FSH in GnRH-AntagoniST Controlled Ovarian Hyperstimulation Cycles (FAST)
Acronym: FAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13EU/FSH01
Record Dates: First submitted 2013-10-08; First posted 2013-10-25 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: In vitro fertilization (IVF); Assisted reproduction technologies (ART); GnRH-antagonist; Follicle stimulating hormone (FSH)
MeSH Terms: conditions — Infertility | interventions — Urofollitropin; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fostimon® (Experimental): 75 IU/vial, powder and solvent for solution for subcutaneous injection (Follicle Stimulating Hormone,IBSA Institut Biochimique SA)
  Interventions: Drug: Urofollitrophin
- Gonal-F® (Active Comparator): 75 IU/vial powder and solvent for solution for subcutaneous injection (Follicle Stimulating Hormone; Merck Serono)
  Interventions: Drug: Follitrophin alpha

INTERVENTIONS:
Drug: Urofollitrophin
  Other Names: human derived follicle stimulation hormone
  Arms: Fostimon®
Drug: Follitrophin alpha
  Other Names: Recombinant follicle stimulation hormone
  Arms: Gonal-F®

SUMMARY:
The purpose of the non-inferiority study is to evaluate the clinical efficacy and the safety of two different subcutaneous FSH preparations (Fostimon versus Gonal-F) for controlled ovarian hyperstimulation in a GnRH-antagonist cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-38 years old;
* BMI: 18-28 kg/m2;
* Less than 3 previously completed IVF cycles;
* Basal FSH <10 IU/L and E2 <80 pg/ml;
* TSH < 2.5 mIU/L
* >10 and <30 antral follicles 2-10 mm in size for both ovaries combined
* AMH: >1 ng/ml (7.15 pmol/l) and <5.6 ng/ml (40.0 pmol/l)
* Presence and adequate visualization of both ovaries;
* Within 12 months of the beginning of the study, uterine cavity consistent with expected normal function as assessed through transvaginal ultrasound, hysterosalpingogram, sonohysterogram or hysteroscopic examination;

Exclusion Criteria:

* Primary ovarian failure or women known as poor responders;
* PCO and PCOS;
* Severe OHSS in a previous COH cycle;
* Uterine malformation that may impair the possibility to get pregnant;
* Ovarian cysts >10 mm;
* Hydrosalpinx that have not been surgically removed or ligated;
* Endometriosis stage 3 or 4;
* Oocyte donation;
* Severe male factor;
* Pathologies associated with any contraindication of being pregnant;
* History of recurrent miscarriage (more than 3 previous miscarriages);
* Hypersensitivity to the study medication;
* Abnormal bleeding of undetermined origin;
* Uncontrolled thyroid or adrenal dysfunction;
* Neoplasias;
* Severe impairment of renal and/or hepatic function.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 710 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Barri, MD, Study Chair — Institut Universitari Dexeus, Barcelona, Spain; Christophe Blockeel, MD, Study Chair — Universitair Ziekenhuis Brussel, Belgium
Locations (16):
- Belgium (2):
  - UCL- Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
- Italy (5):
  - Spedali Civili di Brescia, Brescia
  - Fondazione Ca'Granda, Osp Maggiore Policlinico, Milan
  - IRCCS San Raffaele, Milan
  - Università degli Studi di Napoli 'Federico II', Naples
  - Azienda Ospedaliera Di Reggio Emilia, Reggio Emilia
- Spain (4):
  - Clinica IVI Alicante, Alicante
  - Institut Universitari Dexeus, Barcelona
  - Ginefiv Clínica de Fertilidad, Madrid
  - Instituto Valenciano de Infertilidad (IVI), Seville
- Switzerland (2):
  - Universitäts-Frauenklinik, Basel, Canton of Basel-City
  - Universitätsklinik für Frauenheilkunde, Bern, Canton of Bern
- Turkey (Türkiye) (2):
  - Prof. Bülent Urman, Istanbul
  - Ege University, Izmir
- Midland Fertility Services, Aldridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fostimon®: 75 IU/vial, powder and solvent for solution for subcutaneous injection (Follicle Stimulating Hormone,IBSA Institut Biochimique SA)
  Urofollitrophin
- Gonal-F®: 75 IU/vial powder and solvent for solution for subcutaneous injection (Follicle Stimulating Hormone; Merck Serono)
  Follitrophin alpha
Period: Overall Study
Arm/Group | Fostimon® | Gonal-F®
Started | 352 | 358
Completed | 307 | 313
Not Completed | 45 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostimon® | Gonal-F® | Total
Number analyzed (Participants) | 352 | 358 | 710
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.39 (3.83) | 32.68 (3.52) | 32.53 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 352 | 358 | 710
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 336 | 339 | 675
  Race: Black | 2 | 5 | 7
  Race: Asian | 13 | 14 | 27
  Race: American Indian or Alaska native | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Turkey | 55 | 59 | 114
  Belgium | 39 | 41 | 80
  United Kingdom | 44 | 44 | 88
  Italy | 91 | 88 | 179
  Switzerland | 24 | 25 | 49
  Spain | 99 | 101 | 200

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate
Description: A clinical pregnancy is defined as a pregnancy showing ultrasound embryonic heart activity at 8 weeks of gestation;
Time Frame: 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 352 | 358
percentage of participants | 36.93 | 39.66
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Non-Inferiority — The non-inferiority was evaluated by calculating the 95% CI for the differences in pregnancy rates between the two treatment groups. If the lower bound of the 95% CI of the difference between the two proportions was greater than -0.10 (i.e. 10%), then Fostimon was to be considered not inferior to the control treatment; p = 0.49, Fisher Exact; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-9.88 to 4.42]

2. Secondary Outcome: Number of Follicles >16 mm on the Day of hCG Injection
Time Frame: 10-15 days after starting FSH stimulation
Population: Subject with available data.
Measure: Mean (Standard Deviation); unit: follicles >16 mm
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 347 | 350
follicles >16 mm | 4.10 (2.47) | 4.47 (2.33)
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Number of Oocytes Retrieved
Time Frame: end of treatment period, approximately 2 - 3 weeks.
Population: subjects who underwent oocytes retrieval
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 337 | 346
oocytes | 8.45 (4.72) | 9.33 (4.90)
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.02, ANOVA

4. Secondary Outcome: Fertilization Rate
Time Frame: end of treatment period, approximately 2 - 3 weeks
Population: subjects with at least one oocyte inseminated.
Measure: Mean (Standard Deviation); unit: percentage of oocytes
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 331 | 338
percentage of oocytes | 73.98 (26.44) | 75.85 (21.48)
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.32, ANOVA

5. Secondary Outcome: Embryo Quality (Number of Top Quality Embryos Transferred Per Patient)
Description: The embryo quality evaluation will be performed on culture day 3, just before embryo transfer and will consist in the assessment of blastomeres number and 2 embryo morphology parameters: degree of fragmentation and cell division aspect.
Time Frame: On culture day 3
Population: Subject with at least one embryo transferred, with embryo scoring available.
Measure: Mean (Standard Deviation); unit: Top embryos
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 304 | 314
Top embryos | 0.47 (0.64) | 0.48 (0.64)
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.89, ANOVA

6. Secondary Outcome: Positive Serum Pregnancy Test Rate
Description: Two weeks after embryo transfer, a serum pregnancy test will be performed.
Time Frame: 2 weeks after embryo transfer
Measure: Number; unit: percentage of participants
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 352 | 358
percentage of participants | 47.2 | 49.7
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.5, Fisher Exact

7. Secondary Outcome: Delivery Rate
Time Frame: 9 months
Population: For 4 patients, 3 allocated to the Fostimon® group and 1 allocated to the Gonal-F® group this information was not available because of lost to follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 349 | 357
percentage of participants | 34.4 | 36.7
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.53, Fisher Exact

8. Secondary Outcome: Cumulative Pregnancy Rate
Description: Patients who will not get pregnant during the study, will be allowed to perform a frozen embryo transfer. Cumulative pregnancy rate will include also pregnancies achieved after a frozen embryo transfer.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Fostimon® | Gonal-F®
Number analyzed (Participants) | 352 | 358
percentage of participants | 45.2 | 52.0
Statistical Analysis 1: Comparison: Fostimon® vs Gonal-F®; Test type: Other; p = 0.07, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the signature of the informed consent to the end-of-trial (i.e. up to 9 months in case of a positive pregnancy).
Arm/Group | Fostimon® | Gonal-F®
All-Cause Mortality (participants affected / at risk) | 0/352 | 0/358
Serious Adverse Events (participants affected / at risk) | 24/352 | 31/358
Other Adverse Events (participants affected / at risk) | 36/352 | 42/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostimon® (N=352) | Gonal-F® (N=358)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abortion early (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
imminent abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Multiple pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Oligohydramniosis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Placenta praevia haemorrage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Postpartum haemorrage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
premature delivery (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 7 (7)
premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
intra abdominal haemorrage (Gastrointestinal disorders) | 0 (0) | 1 (1)
peritoneal haemorrage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 (2) | 4 (4)
pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fostimon® (N=352) | Gonal-F® (N=358)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 8 (8)
Headache (Nervous system disorders) | 7 (7) | 11 (15)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 15 (15) | 15 (15)
Vaginal haemorrage (Reproductive system and breast disorders) | 7 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No